CLINICAL TRIAL: NCT04017936
Title: Interleukin-1 Blockade for Treatment of Cardiac Sarcoidosis
Acronym: MAGiC-ART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20015843; R21TR003103 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Sarcoidosis
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Anakinra (Experimental): 100 mg/0.67 mL daily subcutaneous injection for 4 weeks
  Interventions: Drug: Anakinra
- Standard of Care (No Intervention): Continue standard of care treatment

INTERVENTIONS:
Drug: Anakinra — Active Treatment
  Arms: Anakinra

SUMMARY:
Sarcoidosis is a heterogeneous disorder of unknown etiology whose signature lesions are granulomatous inflammatory infiltrates in involved tissues. Tissue commonly affected are lungs, skin, eyes, lymph nodes and the heart. In this latter case, cardiac sarcoidosis (CS) can lead to atrioventricular (AV) blocks, ventricular arrhythmias, heart failure (HF) and sudden cardiac death. Similar to other involved organs, cardiac disease generally progresses from areas of focal inflammation to scar. However, the natural history of CS is not well characterized complicating an immediate and definitive diagnosis. The management of CS often requires multidisciplinary care teams and is challenged by data limited to small observational studies and from the high likelihood of side effects of most of the treatments currently used (eg: corticosteroids, methotrexate and TNF-alfa inhibitors).

Interleukin-1 (IL-1) is the prototypical pro-inflammatory cytokine, also referred to as master regulator of the inflammatory response, involved in virtually every acute process. There is evidence that IL-1 plays a role in mouse model of sarcoidosis and human pulmonary lesions as the presence of the inflammasome in granulomas of the heart of patients with cardiac sarcoidosis, providing additional support for a role of IL-1 in the pathogenesis of CS. However, IL-1 blockade has never been evaluated as a potential therapeutic agent for cardiac sarcoidosis.

In the current study, researchers aim to evaluate the safety and efficacy of IL-1 blockade with anakinra (IL-1 receptor antagonist) in patients with cardiac sarcoidosis.

DETAILED DESCRIPTION:
Researchers will perform an open label randomized clinical trial of anakinra (recombinant IL-1 receptor antagonist, Kineret, SOBI, Sweden) given for 4 weeks in 28 patients with cardiac sarcoidosis (defined using Heart Rhythm Society diagnostic criteria).

ELIGIBILITY:
INCLUSION CRITERIA (all 3 criteria need to be met)

* Clinical diagnosis of cardiac sarcoidosis according to the Heart Rhythm Society or the New Japanese Cardiac Sarcoidosis Guidelines (must meet one of the diagnostic pathways)
* Heart Rhythm Society Diagnostic Criteria based on 2 diagnostic pathways:

  1. Histological diagnosis from myocardial tissue - cardiac sarcoidosis is diagnosed in the presence of non-caseating granuloma on histologic examination of myocardial tissue with no alternative cause identified (including negative stain for microorganisms - as applicable);
  2. Clinical diagnosis from invasive and/or non-invasive studies - it is probable that there is cardiac sarcoidosis if there is (a) histological diagnosis of extracardiac sarcoidosis and (b) one or more of the following: steroid +/- immunosuppressant responsive cardiomyopathy or heart block; unexplained reduction in LVEF (<40%); unexplained sustained (spontaneous or induced) ventricular tachycardia; Mobitz type II 2nd degree or 3rd degree AV block; patchy uptake on dedicated cardiac PET (in a pattern consistent with cardiac sarcoidosis); late gadolinium enhancement on cardiac magnetic resonance (in a pattern consistent with cardiac sarcoidosis); positive gallium uptake (in a pattern consistent with cardiac sarcoidosis) and (c) other causes for the cardiac manifestation(s) have been reasonable excluded.
* Japanese Cardiac Sarcoidosis Diagnostic Criteria:

  1. Histological diagnosis group (those with positive myocardial biopsy findings) Cardiac sarcoidosis is diagnosed histologically when endomyocardial biopsy or surgical specimens demonstrate non-caseating epithelioid granulomas.
  2. Clinical diagnosis group (those with negative myocardial biopsy findings or those not undergoing myocardial biopsy)

The patient is clinically diagnosed as having sarcoidosis:

1. When epithelioid granulomas are found in organs other than the heart and clinical findings strongly suggestive of the above-mentioned cardiac involvement are present (Table 1); or
2. When the patient shows clinical findings strongly suggestive of pulmonary or ophthalmic sarcoidosis; at least 2 of the 5 characteristic laboratory findings of a sarcoidosis (Table 2); and clinical findings strongly suggest the above-mentioned cardiac involvement (Table 1)

TABLE 1. Clinical findings defining cardiac involvement Cardiac findings should be assess based on the major criteria and the minor criteria. Clinical findings that satisfy the following 1) or 2) strongly suggest the presence of cardiac involvement.

1. 2 or more of the 5 major criteria (a)-(e) are satisfied.
2. 1 of the 5 major criteria (a)-(e) and 2 or more of the 3 minor criteria (f)-(h) are satisfied.

1. Major criteria

1. High-grade AV block (including complete AV block) or fatal ventricular arrhythmia (e.g., sustained VT and VF)
2. Basal thinning of the ventricular septum or abnormal ventricular wall anatomy (ventricular aneurysm, thinning of the middle or upper ventricular septum, regional wall thickening
3. Left ventricular contractile dysfunction (LVEF < 50%)
4. 67Ga citrate scintigraphy or 18F-FDG PET reveals abnormally high tracer accumulation in the heart
5. Gadolinium-enhanced MRI revealed delayed contrast enhancement of the myocardium 2. Minor criteria
6. Abnormal ECG findings: Ventricular arrhythmias (nonsustained VT, multifocal or frequent premature ventricular contractions, bundle branch block, axis deviation, or abnormal Q waves
7. Perfusion defects on myocardial perfusion scintigraphy (SPECT)
8. Endomyocardial biopsy: Monocyte infiltration and moderate or severe myocardial interstitial fibrosis

Table 2. Characteristic laboratory findings of sarcoidosis 6. Bilateral hilar lymphadenopathy 7. High serum angiotensin-converting (ACE) activity or elevated serum lysozyme levels 8. High serum soluble interleukin-2 receptor (sIL-2R) levels 9. Significant tracer accumulation in 67Ga citrate scintigraphy or 18F-FDG PET 10. A high percentage of lymphocytes with a CD4CD8 ration of >3.5 in BAL fluid. 11.

* Diagnostic guidelines for isolated cardiac sarcoidosis based on New CS Guidelines in Japan Prerequisite

  1. No clinical findings characteristic of sarcoidosis are observed in any organs other than the heart. (The patient should be examined in detail for respiratory, ophthalmic, and skin involvement of sarcoidosis. When the patient is symptomatic, other etiologies that can affect the corresponding organs must be ruled out.)
  2. 67Ga scintigraphy or 18F-FDG PET reveals no abnormal tracer accumulation in any organs other than the heart.
  3. A chest CT scan reveals no shadow along the lymphatic tracts in the lungs or no hilar and mediastinal lymphadenopathy (minor axis>10 mm).

  <!-- -->

  1. Histological diagnosis group Isolated cardiac sarcoidosis is diagnosed histologically when endomyocardial biopsy or surgical specimens demonstrate non-caseating epithelioid granulomas.
  2. Clinical diagnosis group Isolated cardiac sarcoidosis is diagnosed clinically when criterion (d) and at least 3 other major criteria (a)-(e) are satisfied. (Table 1)
* Cardiac fluoro-deoxyglucose uptake on recent PET (performed within the prior month).
* CRP high-sensitivty assay >2 mg/l.

EXCLUSION CRITERIA (any of the following criteria would result in exclusion)

1. Age<21 years;
2. Pregnancy;
3. Inability to obtain consent from patient or legally authorized representative;
4. Contraindications to treatment with Anakinra (Kineret)(i.e. prior allergic reaction to the drug or to E. coli derived products or severe allergy to latex);
5. Severe anemia (Hgb<8 g/dl - due to the need of more frequent blood sampling with this study).
6. Acute or chronic active infections (not including treated/cured HCV with negative viral load).
7. Acute or chronic inflammatory disease or immunosuppressive therapies (excluding stable [>1 month] oral corticosteroids at a dose of prednisone less than 0.5 mg/kg/day or methotrexate).
8. Active acute or chronic psychiatric illness that in the opinion of the investigator may prevent from complying with study instructions;
9. Limited English Proficiency that in the opinion of the investigator may prevent from understanding the content of the informed consent form or safely completing the study procedures.
10. Live vaccination within the prior month
11. Neutropenia (defined as absolute neutrophil count < 1,500/ml or <1,000/ml if subject is African American)
12. History of malignancy within the prior 5 years (with exception of basal cell skin cancer, carcinoma in-situ of the cervix or low risk prostate cancer after curative therapy)
13. Participation in another concurrent intervention study within 30 day or treatment with an investigational drug within 5 half-lives prior to randomization
14. Severe kidney disease (GFR <30 mL/min/1.73m2)
15. Evidence of COVID-19 within the last 60 days or recent (21 days) exposure to close personal contact with COVID-19.
16. [Chronic, moderate-to-severe kidney disease (GFR <60 mL/min/1.73m2) or acute kidney injury, or history of severe hypersensitivity reactions to gadolinium-based contrast agents] - For VCU Imaging Substudy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Kron, MD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - University of Michigan Sarcoidosis Clinic, Ann Arbor, Michigan
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kron J, Crawford T, Bogun F, Jordan JH, Koelling T, Syed H, Syed A, Iden T, Polly K, Federmann EG, Bray K, Lathkar-Pradhan S, Ladd A, Dickson VM, Barron A, Tavoosi A, Beanlands R, Birnie D, Ellenbogen K, Van Tassell BW, Gregory Hundley W, Abbate A. Interleukin-1 Blockade in Cardiac Sarcoidosis: A Pilot Study. Circ Arrhythm Electrophysiol. 2023 May;16(5):e011869. doi: 10.1161/CIRCEP.123.011869. Epub 2023 Apr 24. No abstract available. PMID 37092332
- [Derived] Kron J, Crawford T, Mihalick V, Bogun F, Jordan JH, Koelling T, Syed H, Syed A, Iden T, Polly K, Federmann E, Bray K, Lathkar-Pradhan S, Jasti S, Rosenfeld L, Birnie D, Smallfield M, Kang L, Fowler AB, Ladd A, Ellenbogen K, Van Tassell B, Gregory Hundley W, Abbate A. Interleukin-1 blockade in cardiac sarcoidosis: study design of the multimodality assessment of granulomas in cardiac sarcoidosis: Anakinra Randomized Trial (MAGiC-ART). J Transl Med. 2021 Nov 8;19(1):460. doi: 10.1186/s12967-021-03130-8. PMID 34749739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra | Standard of Care
Started | 7 | 10
Completed | 7 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra | Standard of Care | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [53 to 64] | 61 [48 to 64] | 61 [48 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammation Marker
Description: Change in c-reactive protein in participant plasma samples
Time Frame: Baseline to 28 days
Population: Patient 5 excluded from Anakinra group outcome analysis.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Anakinra | Standard of Care
Number analyzed (Participants) | 6 | 10
mg/L | -43 (36) | 7 (41.56)

2. Secondary Outcome: Change in Cardiac Fibrosis
Description: Change in late gadolinium enhancement evident on magnetic resonance imaging (MRI) scan
Time Frame: Baseline to 180 days
Population: Reported as percent change of relative enhanced late gadolinium enhancement volume (%)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Anakinra | Standard of Care
Number analyzed (Participants) | 2 | 3
percentage change | 17.7 (14.7) | 12.3 (13.3)

ADVERSE EVENTS:
Time Frame: 180 days
Description: Regular investigator assessment, phone call follow-up.
Arm/Group | Anakinra | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/10
Other Adverse Events (participants affected / at risk) | 7/7 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=7) | Standard of Care (N=10)
hospitalized for a diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=7) | Standard of Care (N=10)
Serious Infection (Infections and infestations) | 1 (1) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Recurrent atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Rhinovirus (Infections and infestations) | 1 (1) | 0 (0)
Abdominal fullness (Infections and infestations) | 1 (1) | 1 (1)
Worsening kidney function (Infections and infestations) | 1 (1) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypermatabolic lymph nodes (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Skin Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT04017936/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04017936/ICF_001.pdf